CLINICAL TRIAL: NCT02849821
Title: A Study on the Influence of Hypoxia on Healthy Volunteers and Patients With Inflammatory Bowel Disease (IBD): The Altitude IBD Study
Brief Title: The Altitude Inflammatory Bowel Disease Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: Triemli Hospital (Other); Zurich Center for Integrative Human Physiology (Other); Institute of Biostatistics (Unknown); Insel Gruppe AG, University Hospital Bern (Other); Institute of Physiology Irchel (Unknown); Institute of Veterinary Physiology (Unknown); Swiss Aeromedical Center Switzerland (Unknown); Institute of Experimental Immunology (Unknown); University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: VAV003
Record Dates: First submitted 2016-07-12; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Sigmoidoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hypobaric pressure chamber (Other): The healthy volunteers and IBD patients will have a 3-hour exposure to hypoxic conditions simulating an altitude of 4,000 meters above sea level (m.a.s.l.) in a hypobaric pressure chamber. Before and after the pressure chamber sigmoidoscopy will be performed. During stay in the pressure chamber repetitive measurements of bladder volume will be performed by sonography.
  Interventions: Other: hypobaric pressure chamber; Other: Sigmoidoscopy

INTERVENTIONS:
Other: hypobaric pressure chamber — hypobaric chamber: ascent within 10 minutes, 3 hour exposure to hypoxic conditions simulating an altitude of 4,000 m.a.s.l., afterwards controlled descent under continuous pulsoximetric control
Other: Sigmoidoscopy — To retrieve biopsies from the colon during the course of the study 3 sigmoidoscopies were performed. The first sigmoidoscopy was performed 1 day before the stay in the hypobaric chamber. The second sigmoidoscopy was performed directly after the hypobaric chamber and the third sigmoidoscopy was performed 1 week after the hypobaric chamber. During each sigmoidoscopy 6 biopsies were taken with standard size forceps (2.4 mm). One biopsy was analysed by real-time quantitative polymerase chain reaction (PCR), one biopsy was analysed by Western blotting and another biopsy was analysed for gene gene-expression by in situ hybridisation. Two biopsies were analysed by immunohistochemistry (IHC) and one biopsy was stained with hematoxylin and eosin (H&E).

SUMMARY:
This is a prospective, controlled and observational study. Participants underwent a 3-hour exposure to hypoxic conditions simulating an altitude of 4,000 meters above sea level (m.a.s.l.) in a hypobaric pressure chamber. Clinical parameters, as well as blood and stool samples and biopsies from the sigmoid colon (by sigmoidoscopy) are collected at subsequent time points. The investigators goal is to evaluate if a 3-hour stay at high altitude (4, 000 m) can alter disease activity and can modulate a pro inflammatory reaction.

DETAILED DESCRIPTION:
To evaluate the potential influence of hypoxia on the course of IBD on a biomolecular level, and to test the effects of hypoxia under standardized conditions, the investigators initiated a prospective and controlled investigation in healthy controls and IBD patients in stable remission. the investigators primary aim is to show that a 3-hour stay at high altitude can alter disease activity of IBD. Ten healthy volunteers, 11 Crohn's disease (CD) patients and 9 ulcerative colitis (UC) patients underwent a 3-hour exposure to hypoxic conditions simulating an altitude of 4,000 m.a.s.l. in a hypobaric low-pressure chamber situated at the Swiss Aeromedical Center, Dubendorf, Switzerland. Stool samples for the analysis of calprotectin and microbiotal composition, biopsy samples from the rectosigmoid region, and blood samples were repetitively collected and analysed in conjunction with detailed records of clinical symptoms over a subsequent interval of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* had a diagnosis of Crohn's disease or ulcerative colitis at least 6 months prior to inclusion
* gave written consent
* were in clinical remission (measured by Harvey Bradshaw Activity Index (HBI) in CD and the partial Mayo Score for UC)

Exclusion Criteria:

* had contraindications for a sigmoidoscopy
* had intercurrent bacterial or viral intestinal disease (by culture or serology)
* were pregnant or breast feeding
* had a severe concomitant disease which excluded from participating in the study by means of the study physician
* were likely to or showed no cooperation for the study procedures
* had active infection or systemic antibiotic, antiviral or antifungal treatment 3 weeks before baseline
* were suffering from short-bowel syndrome
* were receiving parenteral nutrition
* had a clinical condition which did not allow a stay at heights of 4,000 m.a.s.l.
* were claustrophobic

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change of Harvey Bradshaw Activity Index (HBI) | 4 weeks
  Harvey Bradshaw Activity Index (HBI) in Crohn's disease (CD):
  To calculate the clinical activity of patients with CD the Harvey Bradshaw Activity Index (HBI) was used. This index includes general wellbeing, abdominal pain, the number of bowel movements, abdominal resistance and CD associated extraintestinal diseases. Each category has a point value assigned and from the sum of all categories a point value is calculated.
Change of partial Mayo Score | 4 weeks
  partial Mayo Score for Ulcerative Colitis (UC): To calculate the clinical activity of patients with UC the partial Mayo Score was used. This clinical index includes the stool frequency, the amount of blood in the stool and the physician rating of disease activity. Each category has a point value assigned from 0 to 3 and from the sum of all categories a point value was calculated. Remission is defined as 0-1 points, mild disease 2-4 points, moderate disease 5-6 points and severe disease as 7-9 points.

SECONDARY OUTCOMES:
change in levels of hypoxia-inducible factor (HIF)-1 | 4 weeks
Change in bladder volume | 4 weeks
  measured by sonography (ml)
Change in levels of angiotensin and vasopressin in urine | 4 weeks
Change in levels of catecholamines (adrenaline and noradrenaline) in blood | 4 weeks
Change in pro- and anti-inflammatory cytokins | 4 weeks
  tumor necrosis factor alpha (TNF-α), tumor necrosis factor (TNF), interleukin-1β (IL-1β), interferon-gamma (IFNg), interleukin-10 (IL-10)
Inflammation in sigmoid colon | 4 weeks
  Assessed by sigmoidoscopy:
  signs of inflammation:
  * decreased vascular pattern
  * ulcers
  * bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Stephan R Vavricka, Prof. Dr., Principal Investigator — University of Zurich

REFERENCES:
- [Derived] Vavricka SR, Zeitz J, Madanchi M, Ruiz PA, Biedermann L, Morsy Y, Yilmaz B, Scharl M, Scharl S, Gassmann M, Lutz TA, Kunz A, Bron D, Misselwitz B, MacPherson AJ, Rogler G, Greuter T. A Prospective Interventional Study to Evaluate the Effect of Hypoxia on Healthy Volunteers and Patients With Inflammatory Bowel Disease: The Altitude Inflammatory Bowel Disease Study. Am J Gastroenterol. 2025 Dec 16. doi: 10.14309/ajg.0000000000003888. Online ahead of print. PMID 41400272
- [Derived] Vavricka S, Ruiz PA, Scharl S, Biedermann L, Scharl M, de Valliere C, Lundby C, Wenger RH, Held L, Merz TM, Gassmann M, Lutz T, Kunz A, Bron D, Fontana A, Strauss L, Weber A, Fried M, Rogler G, Zeitz J. Protocol for a prospective, controlled, observational study to evaluate the influence of hypoxia on healthy volunteers and patients with inflammatory bowel disease: the Altitude IBD Study. BMJ Open. 2017 Jan 5;7(1):e013477. doi: 10.1136/bmjopen-2016-013477. PMID 28057654